CLINICAL TRIAL: NCT00142701
Title: Enhancing Support for Women at Risk for Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 251; R01HL062156 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Coronary Heart Disease Risk Reduction; Diabetes Mellitus, Non-insulin Dependent
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Diabetes Mellitus, Type 2 | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: diet
Behavioral: physical activity
Behavioral: stress management
Behavioral: smoking cessation

SUMMARY:
To test a practical, theory-based intervention to achieve long-term behavior change for postmenopausal women with Type 2 diabetes at high risk for developing coronary heart disease (CHD).

DETAILED DESCRIPTION:
BACKGROUND:

The overall goal of this study was to test a practical, theory-based intervention to achieve long-term behavior change for women with Type 2 diabetes at high risk for developing coronary heart disease (CHD). Epidemiological and clinical studies suggest that diabetes is associated with increased risk for CHD that is greater in women than in men. CHD is a major cause of death and functional limitations in women, but the vast majority of CHD studies have primarily involved middle-aged men. There is convincing research evidence that healthy lifestyle behaviors, including low-fat diet, physical activity, stress management, smoking cessation, and social support, can reduce CHD risk

The study was initiated in response to a Request for Applications released in October 1997 by the National Institutes of Health Office of the Director on "Innovative Approaches to Disease Prevention Through Behavior Change."

DESIGN NARRATIVE:

The study was a randomized trial to compare short-term (6-month) outcomes in women receiving usual care compared to a modified Ornish-type comprehensive lifestyle management (CLM) intervention. Participants (N = 279) were randomized to usual care (UC) or Mediterranean Lifestyle Program, a lifestyle change intervention aimed at the behavioral risk factors (eating patterns, physical activity, stress management, and social support) affecting risk for CHD in postmenopausal women with type 2 diabetes. After 6 months, women in the CLM condition were randomized to one of two approaches for providing support either lay-led group support or personalized computer-based support - to evaluate these strategies in enhancing longer-term maintenance of effects. Outcomes included multiple CHD lifestyle behaviors (e.g., dietary intake, exercise levels, stress management, smoking cessation), physiological risk factors associated with CHD (e.g., serum lipids, hypertension, weight, vascular reactivity), HbA1c (glycated hemoglobin, a measure of diabetes), and quality of life (e.g., depression, functioning).

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-04; Primary Completion 2004-09 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Toobert — Oregon Research Institute

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toobert DJ, Strycker LA, Glasgow RE, Barrera M Jr, Angell K. Effects of the mediterranean lifestyle program on multiple risk behaviors and psychosocial outcomes among women at risk for heart disease. Ann Behav Med. 2005 Apr;29(2):128-37. doi: 10.1207/s15324796abm2902_7. PMID 15823786
- [Background] Glasgow RE, Toobert DJ, Barrera M Jr, Strycker LA. The Chronic Illness Resources Survey: cross-validation and sensitivity to intervention. Health Educ Res. 2005 Aug;20(4):402-9. doi: 10.1093/her/cyg140. Epub 2004 Nov 30. PMID 15572438
- [Background] Toobert DJ, Glasgow RE, Strycker LA, Barrera M Jr, Radcliffe JL, Wander RC, Bagdade JD. Biologic and quality-of-life outcomes from the Mediterranean Lifestyle Program: a randomized clinical trial. Diabetes Care. 2003 Aug;26(8):2288-93. doi: 10.2337/diacare.26.8.2288. PMID 12882850
- [Background] Toobert DJ, Strycker LA, Glasgow RE, Barrera M, Bagdade JD. Enhancing support for health behavior change among women at risk for heart disease: the Mediterranean Lifestyle Trial. Health Educ Res. 2002 Oct;17(5):574-85. doi: 10.1093/her/17.5.574. PMID 12408202
- [Background] Toobert DJ, Strycker LA, Glasgow RE, Bagdade JD. If you build it, will they come?. Reach and Adoption associated with a comprehensive lifestyle management program for women with type 2 diabetes. Patient Educ Couns. 2002 Oct-Nov;48(2):99-105. doi: 10.1016/s0738-3991(02)00120-9. PMID 12401412